CLINICAL TRIAL: NCT06169228
Title: Impact of Treatment With Mandibular Advancement Device (MAD) on Sleep Quality in Patients With Obstructive Sleep Apnea (OSA)
Brief Title: Mandibular Advancement Device on Sleep Quality in Obstructive Sleep Apnea Patients
Acronym: DAMOSA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Principal Investigator, Maria Fernanda Troncoso, Investigador principal, Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz
Other Study IDs: PI19/00830
Record Dates: First submitted 2023-01-30; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Mandibular Advancement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

INTERVENTIONS:
Device: mandibular advancement — The multidisciplinary sleep unit assessment and follow-up protocol will be followed for this group of patients based on the Spanish Clinical Practice Guideline of the Spanish Sleep Society (SES) on the use of mandibular advancement devices in the treatment of patients with obstructive sleep apnea

SUMMARY:
Sleep is an important factor that influences long-term quality of life with known health consequences. Obstructive sleep apnea, the most prevalent disease that disturbs sleep, is considered a public health problem. Treatment with continuous positive airway pressure is cost effective and reverses the clinical consequences but there is a percentage of patients who do not tolerate it or leave it without treatment and with potential future health complications. Mandibular advancement device can be a valid and well tolerated alternative, it is known that it reduces apnea-hypopnea index, but its effect on the improvement of sleep quality is evaluated by polysomnography that interferes with the quality of sleep. There is an ambulatory monitoring device for sleep quality and circadian rhythms, which can register prolonged periods of time, under natural conditions and at a lower cost than a polysomnography. This pilot project assesses whether mandibular advancement device is an effective and well tolerated alternative in the treatment of obstructive sleep apnea to improve the quality of life and sleep in the medium and long term.

DETAILED DESCRIPTION:
Design: observational, unicentric prospective. 50 patients / year will be included, for 3 years. The care protocol (evaluation and follow-up) of the multidisciplinary sleep unit will be followed. Demographic and anthropometric data will be collected. The dental status of the temporo-mandibular joint will be assessed. Radiological records, home respiratory polygraphy, ambulatory monitoring device for 7 days , quality of life questionnaires before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Obstructive Sleep Apnea Syndrome
* opt for mandibular advancement device as 1st treatment alternative
* opt for mandibular advancement device due to intolerance to continuous positive airway pressure

Exclusion Criteria:

* Patient with orthodontics, malocclusion and periodontal or temporomandibular joint disease who, after assessment by dentistry contraindicates it.
* Central Sleep apnea (more than 50% of central events in the baseline polygraph).
* Under 18 years old.
* Pregnancy
* Comorbidities that can potentially alter sleep architecture.
* Psychophysical inability to complete questionnaires.
* Not obtaining informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who come to the Multidisciplinary sleep unit of the Fundación Jiménez Díaz with suspicion of Obstructive sleep apnea and who present an Apnea Hypopnea Index greater than five
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
mandibular advancement device on sleep quality | 3 years
  Tolerability and efficacy of treatment with a mandibular advancement device (MAD) on sleep quality in patients with Obstructive Sleep Apnea (OSA) measured by the ambulatory circadian monitoring device.
ambulatory circadian monitoring device | 3 years
  To evaluate improvement in sleep quality with mandibular advancement devices measured by fragmentation and stability of sleep by the circadian monitoring sensor.
home sleep apnea test | 3 years
  To evaluate the number of residual apneic breaths measured by home home sleep apnea test

SECONDARY OUTCOMES:
Obstructive sleep apnea severity | 3 years
  Evaluate the severity by home sleep apnea test
questionnaire SF-12 | 3 years
  multidimensional health related quality of life
questionnaire EuroQoL | 3 years
  standardized non-disease specific instrument to describe and value health-related quality of life
questionnaire iPAQ | 3 years
  International Physical Activity Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Maria Fernanda Troncoso Acevedo, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No